CLINICAL TRIAL: NCT06055842
Title: Retrospective Study on the Effect of Different Implant Positions for Implant Retained Mandibular Overdenture: Radiographic Evaluation of the Circumferential Bone Level and Bone Remodeling in the Anterior and Posterior Mandible
Brief Title: Different Implant Positions for Implant Retained Mandibular Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Khloud Ezzat, lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M0108023RP
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2023-09

CONDITIONS: Bone Loss
Keywords: implant; overdenture
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Denture, Overlay

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lateral incisor group (Active Comparator): Patients having two mandibular implants in lateral incisor positions.
  Interventions: Other: over-denture
- canine group (Active Comparator): Patients having two mandibular implants in canine positions
  Interventions: Other: over-denture

INTERVENTIONS:
Other: over-denture — implant retained overdenture prosthesis.

SUMMARY:
This study will aim to evaluate the effect of two different implant positions, lateral incisors, and canine areas, on anterior and posterior ridge resorption and bone remodeling after different periods of denture insertion.

DETAILED DESCRIPTION:
Twelve patients will be recruited from a previous study (14), having two-implant mandibular overdentures. Patients recalled from the database set of the clinic of the Removable Prosthodontic Department, Faculty of Dentistry, Mansoura University. The patients will be grouped based on the position of the two implants.

All patients will be informed about all prosthetic procedures that will be done. Also, they will sign the consent form of the ethical committee of the faculty of dentistry, at Mansoura University.

All selected patients with the following criteria: mandibular two implants retained overdenture opposing complete edentulous maxillary arch, attended the previous follow-up recalls with previous CBCT examination. Patients who didn't attend previous follow-up recalls, didn't perform radiographic follow-up, or had para-functional habits will excluded from the study Patients will be divided into two groups Group A (6 patients): Patients having two mandibular implants in lateral incisor positions.

Group B (6 patients): Patients having two mandibular implants in canine positions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular two implants retained overdenture opposing complete edentulous maxillary arch,
* attended the previous follow-up recalls with previous CBCT examination.

Exclusion Criteria:

* Patients who didn't attend previous follow-up recalls, didn't perform radiographic follow-up, or had para-functional habits will be excluded from the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
implant survival rate | 5 years
  index
circumferential bone loss | 5 years
  peri-implant bone changes in mm
posterior bone changes | 5 years
  bone loss in mm

CONTACTS AND LOCATIONS:
Overall Officials: Khloud Ezzat, Principal Investigator — Lecturer
Locations (1):
- Khloud Ezzat, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mourad KE, Emera RMK, Habib A. Effect of different implant positions for two implant-retained mandibular overdenture: a retrospective 5-years radiographic evaluation of the circumferential peri-implant bone loss and posterior ridge resorptive changes. BMC Oral Health. 2024 Sep 30;24(1):1161. doi: 10.1186/s12903-024-04871-w. PMID 39350107